CLINICAL TRIAL: NCT02870153
Title: A Randomized Phase II Study of Oxaliplatin and S-1 (SOX) Versus Oxaliplatin and Capecitabine (XELOX) in Patients With Peritoneal Metastasis of Colorectal Cancer
Brief Title: SOX Versus XELOX for Patients With Peritoneal Metastasis of Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZYY-CRC-007
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; titanium silicide; XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOX(oxalipaltin+S-1) (Experimental): Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days
  Interventions: Drug: SOX
- XELOX (oxalipaltin+capecitabine) (Active Comparator): Oxaliplatin 130mg/m2 IV on D1 every 21 days and Capecitabine 2000mg/m2/day PO, divided by two on D1-14 every 21 days
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: SOX — Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days
  Other Names: Eloxatin; TS-1
  Arms: SOX(oxalipaltin+S-1)
Drug: XELOX — Oxaliplatin 130mg/m2 IV on D1 every 21 days and Capecitabine 2000mg/m2/day PO, divided by two on D1-14 every 21 days
  Other Names: Eloxatin; Xeloda
  Arms: XELOX (oxalipaltin+capecitabine)

SUMMARY:
The aim of this study is to compare the activity and safety of Oxaliplatin and S-1 (SOX) and Oxaliplatin and Capecitabine (XELOX) in patients with peritoneal metastasis of colorectal cancer.

DETAILED DESCRIPTION:
Peritoneal dissemination from colorectal cancer is common, and it has been traditionally regarded as end-stage disease only amenable to palliation by systemic chemotherapy (sCT), or supportive care .Oxaliplatin and oral fluoropyrimidines (capecitabine or S-1) are active agents for colorectal cancer. Recent a phase II trial of combination chemotherapy of oxaliplatin with S-1 (OS) and several phase II trial of combination chemotherapy of oxaliplatin with capecitabine (XELOX) demonstrated good activity and mild toxicity in advanced colorectal cancer. Oxaliplatin and S-1 or capecitabine have distinct mechanisms of action and no overlap of key toxicities. Furthermore, oxaliplatin and fluorouracil were shown to be highly synergistic, not only in preclinical models but also in subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed colorectal adenocarcinoma, initially diagnosed or recurred

Peritoneal metastasis of colorectal cancer

At least one uni-dimensional measurable lesion by RECIST criteria

Age 18 to 80 years old

Estimated life expectancy ≥3 months

ECOG performance status ≤2

Adequate bone marrow function (WBCs ≥ 4,000/µL or absolute neutrophil count ≥ 1,500/µL, platelets ≥ 100,000/µL)

Adequate kidney function (creatinine < 1.5 mg/dL)

Adequate liver function (bilirubin < 2.0 mg/dL, transaminase levels <2.5 times the upper normal limit)

Written informed consent

Exclusion Criteria:

Other tumor type than adenocarcinoma

Previous history of chemotherapy (exception : neoadjuvant or adjuvant chemotherapy without oxaliplatin)

Presence of CNS metastasis, psychosis, or seizure

Obvious bowel obstruction

Evidence of serious gastrointestinal bleeding

Past or concurrent history of neoplasm other than colorectal adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri

Pregnant or lactating women, women of childbearing potential not employing adequate contraception

Other serious illness or medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6 weeks
  According to the RECIST criterion

SECONDARY OUTCOMES:
Side-effect | 8 weeks
  Safety was evaluated according to the NCI-CTC
Time to Progression | 6 years
  According to the RECIST criterion
Overall Survival | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Changping Wu, M.D., Study Director — The First People's Hospital of Changzhou
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Baratti D, Kusamura S, Pietrantonio F, Guaglio M, Niger M, Deraco M. Progress in treatments for colorectal cancer peritoneal metastases during the years 2010-2015. A systematic review. Crit Rev Oncol Hematol. 2016 Apr;100:209-22. doi: 10.1016/j.critrevonc.2016.01.017. Epub 2016 Jan 22. PMID 26867984
- [Background] Esquivel J. Colorectal cancer with peritoneal metastases: Progress, not perfection. J Surg Oncol. 2015 Jul;112(1):115. doi: 10.1002/jso.23954. Epub 2015 Jul 7. No abstract available. PMID 26153356
- [Background] Ogawa M, Anan T, Suzuki T, Okuma M, Ichihara K, Hasegawa T, Yoshida K, Yanaga K. Initial Report of Phase II Study on Bi-weekly SOX plus Cetuximab Treatment for Wild-type K-RAS Advanced and Recurrent Colorectal Cancer. Anticancer Res. 2016 May;36(5):2505-11. PMID 27127165
- [Background] Wang ZQ, Zhang DS, Xu N, Luo DY, Deng YH, Wang FH, Luo HY, Qiu MZ, Li YH, Xu RH. Phase II study of oxaliplatin combined with S-1 and leucovorin (SOL) for Chinese patients with metastatic colorectal cancer. Chin J Cancer. 2016 Jan 6;35:8. doi: 10.1186/s40880-015-0061-3. PMID 26739998